Repetitive position change improves gastric cleanliness for magnetically controlled

capsule gastroscopy

Document Date: May 1, 2018

**Trial registration:** ClinicalTrials.gov, ID: NCT03514966

Yuan-Chen Wang<sup>1,2</sup>, M.D., Jun Pan<sup>1,2</sup>, M.D., Xi Jiang<sup>1,2</sup>, M.D., Xiao-Ju Su<sup>1</sup>, M.D., Wei Zhou<sup>1</sup>,

M.D., Wen-Bin Zou<sup>1</sup>, M.D., Yang-Yang Qian<sup>1</sup>, M.D., Yi-Zhi Chen<sup>1</sup>, M.D., Xiao Liu<sup>1</sup>, M.D., Jin

Yu<sup>1</sup>, M.D., Xiao-Nan Yan<sup>1</sup>, M.D., An-Jing Zhao<sup>1</sup>, M.D., Zhao-Shen Li<sup>1</sup>, M.D., Zhuan Liao<sup>1,\*</sup>,

M.D.

<sup>1</sup>National Clinical Research Center for Digestive Diseases; Department of Gastroenterology,

Changhai Hospital, Second Military Medical University, Shanghai, China

<sup>2</sup>These authors contributed equally to this work

\*Correspondence

Zhuan Liao

National Clinical Research Center for Digestive Diseases; Department of Gastroenterology,

Changhai Hospital, Second Military Medical University, 168 Changhai Road, Shanghai

200433, China

Tel: 86-21-31161004; Fax: 86-21-65492727

E-mail: liaozhuan@smmu.edu.cn

Funding: This study is supported by grants from the National Natural Science Foundation of

China (to Z. Liao, No.81422010); Foundation for the Author of National Excellent Doctoral

Dissertation of China (to Z. Liao, No.201271); the Shuguang Program of Shanghai Education

Development Foundation and Shanghai Municipal Education Commission (to Z. Liao,

No.15SG33); the Chang Jiang Scholars Program of Ministry of Education (to Z. Liao, No.

Q2015190); and Shanghai Sailing Program (to J. Pan, No. 18YF1422800), China.

Author contributions: Study concept and design (ZL); registration of the study (YCW, JP); conduct of the study (YCW, JP); acquisition of data (YCW, XJS, XJ, WBZ, YYQ, WZ, XL, JY, XNY, AJZ); analysis and interpretation of data (YCW, JP); drafting of the manuscript (JP); statistical analysis (YCW); critical revision of the manuscript for important intellectual content (ZL, ZSL); obtained funding (ZL, JP). All authors had access to the study data and reviewed and approved the final manuscript.

Competing Interests: None.

Acknowledgement: None.

## Statistical analysis

In order to define the sample size, we carried out an exploratory study enrolling 20 patients in each group. Mean gastric cleanliness score in the position change and conventional groups were 20.1 and 19.4, respectively. This study was a superiority study based on two-sided alpha as 0.05 and the power as 80%, thus 64 patients (32 patients in each group) were required by using NCSS-PASS 11 program (version 11.0.7, NCSS, Kaysville, Utah, USA). Considering a withdrawal rate of 20%, we enrolled 80 patients at least. Statistical analysis was performed using SPSS Statistics software version 18.0. Descriptive statistics were given as means ± standard deviation (SD). Differences in categorical variables between patient groups were compared by using the Chi-square test; differences in means were compared with the independent *t*-test. In GCS comparison and subgroup analysis which lack of normal distribution for quantitative data, we used Mann-Whitney test for comparison of the two groups. A *P*-value of < 0.05 was considered to be statistically significant.